CLINICAL TRIAL: NCT04198142
Title: Treatment of Nightmares in Psychiatric Inpatients With Imagery Rehearsal Therapy: A Randomized Controlled Trial
Brief Title: Psychiatric Inpatient Nightmare Treatment
Acronym: PINIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00773
Record Dates: First submitted 2019-10-03; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Nightmare; Psychiatric Disorder
Keywords: Psychiatric inpatient care
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagery Rehearsal Therapy Intervention (Experimental): This group receives one to two sessions of Imagery Rehearsal Therapy.
  Interventions: Behavioral: Imagery Rehearsal Therapy
- Treatment as Usual with dream diaries (Active Comparator): This group receives the usual inpatient care without additional Imagery Rehearsal Therapy sessions, but also keeps dream diaries.
  Interventions: Behavioral: Treatment as Usual with dream diaries

INTERVENTIONS:
Behavioral: Imagery Rehearsal Therapy — The Imagery Rehearsal Therapy (IRT) intervention used in this study is a short version of the treatment, consisting of 1-2 sessions.
  The protocol starts with a very brief explanation of the treatment. Then the patient will be guided through an imagery exercise. The next step is to choose a nightmare. This nightmare is then rescripted to a new narrative, which is in no way distressing to the patient anymore. Subsequently, the therapist will guide the patient through an imagery exercise with the new narrative. The new narrative is then either written down or recorded. Lastly, the therapist will explain to the patient, that he or she should rehearse the new narrative daily with imagery exercises.
  Arms: Imagery Rehearsal Therapy Intervention
Behavioral: Treatment as Usual with dream diaries — Treatment as Usual means that patients in this arm will receive usual inpatient care. Additionally, they will keep a dream diary. It has been shown in previous studies that keeping a dream diary has a positive effect on nightmares.
  Arms: Treatment as Usual with dream diaries

SUMMARY:
Nightmares are repeated extremely dysphoric and well-remembered dreams, which typically occur during REM sleep in the second half of sleep, may awaken the dreamer, and upon awakening, individuals quickly become oriented and conscious of their surroundings. Nightmares are very common in psychiatric populations. In psychiatric populations, nightmares can occur as a freestanding disorder, persist in patients after undergoing treatment for a psychiatric disorder, and function as a risk and exacerbating factor regarding psychiatric symptoms. Imagery Rehearsal Therapy (IRT) is a cognitive-behavioral-oriented treatment for nightmares and asks patients to identify an especially distressing nightmare and then works together with the patient on changing the nightmare to a more positive theme, story line, or ending. The new contents are then rehearsed using imagery techniques. IRT is often recommended by guidelines. However, IRT has not been investigated in a randomized controlled trial in the population of psychiatric inpatients. In this study, sixty inpatients with nightmares will be recruited from the inpatient units of the Psychiatric University Hospital Zurich (PUK). Participants will be randomly assigned to an Imagery Rehearsal Therapy (IRT) group or a Treatment As Usual (TAU) control group. Questionnaires and dream diaries will measure changes in nightmare frequency, nightmare distress, nightmare effects, nightmare content, overall sleep quality, dream experiences and believes, symptom severity of primary psychiatric diagnoses, and psychotherapy motivation and hopefulness one week and two weeks after one IRT or TAU session. The TAU group will receive a session in which potential problems with the dream diary will be discussed. Patients in the IRT group will be instructed to use imagery exercises with the new dream narrative for 10 to 15 minutes a day for the duration of the study period.

DETAILED DESCRIPTION:
Nightmares are repeated extremely dysphoric and well-remembered dreams, which typically occur during REM sleep in the second half of sleep (late in the night or during the early morning hours) and upon awakening, individuals quickly become oriented, alert, and conscious of their surroundings. Standard definitions for nightmares often include awakening as an essential criterion, though research suggests that this is not always the case and not all researchers have adopted this waking criterion. Furthermore, although most nightmares occur during REM sleep, they can also occur during non-Rem sleep. Nightmares are very common in psychiatric populations. Studies have found nightmare prevalence rates of 28.4% and 17.5% in depression, 15.6% in anxiety disorders, 24.4% to 25.6% in drug or alcohol abuse, 60% to 90% in Posttraumatic stress disorder (PTSD), and 48% in psychotic disorders. Furthermore, since nightmares often do awaken the individual during the sleep cycle and can make returning to sleep difficult, nightmares can have indirect negative effects through sleep deprivation, which can lead to impaired attention, alertness, reaction time, cognitive processing capacity, memory, mood, ability to stay awake, and heightened pain sensitivity. However, nightmares can also have direct and specific effects. They can affect daily functioning and overall well-being. These implications are even more pronounced in individuals with mental health disorders, where negative outcomes of nightmares were found to often be independent of the co-morbid mental disorders. In psychiatric disorders, nightmares can function as a risk factor, a symptom, and as an exacerbating factor regarding psychiatric symptoms. Nightmares were also found to be significantly associated with higher risk of suicidal ideation, suicide, repeat suicide attempts, and death by suicide, often after controlling for co-morbid mental and other sleep disorders. One cognitive-behavioral-oriented treatment for nightmares is called Imagery Rehearsal Therapy (IRT). IRT asks patients to identify an especially distressing (possibly recurrent) nightmare and works together with the patient on changing the nightmare to a more positive theme, story line, or ending. The new contents are then rehearsed using imagery techniques. In IRT the nightmare can be changed in any way. Some authors argue that imagery rescripting may improve the perceived mastery over nightmares by providing a form of coping by rescripting them. Some authors Arntz speculate that imagery rescripting might modify the fear memory, leading to a reconsolidation with a new meaning that no longer prompts a strong fear response. Imagery rescripting might change the meaning of the original images and the associated automatic emotional processes. Since exposure is not considered to be the most important component of IRT, some authors have pointed out, that the new dream narrative does not have to include material from the original disturbing dream, where solution-oriented thinking may be triggered. IRT is currently among the most studied psychological approaches and is often recommended by guidelines with moderate to large effect sizes. IRT has been shown to be effective for the reduction of nightmare frequency, intensity, and distress. Effects have also been found on depression, anxiety, PTSD symptom severity, sleep quality, insomnia symptoms, and potentially on suicidal ideation. IRT has been used successfully for the treatment of posttraumatic and idiopathic nightmares with sexual assault victims with PTSD, war veterans with PTSD, psychiatric outpatients with various disorders, such as personality disorders, mood disorders, anxiety disorders, and PTSD, and with patients experiencing symptoms of psychosis. Studies have found long-term effects of IRT at follow-ups of 3, 6, 9 and up to 30 months.

To the knowledge of the investigators, there is no randomized controlled trial (RCT), which has investigated the efficacy of IRT in psychiatric inpatients. In order to design the most effective treatment protocol for nightmares, it is necessary to find what works for whom, and how it works. Thus, the proposed project aims to investigate the efficacy of IRT in an RCT with psychiatric inpatients with various disorders. The primary research question is whether IRT has a positive effect on nightmares of psychiatric inpatients in terms of frequency, distress, and intensity, which constitute the outcomes typically used to assess nightmares. A secondary research question is if certain nightmare characteristics and / or treatment characteristics moderate treatment efficacy.

For this study, sixty inpatients with nightmares will be recruited from the inpatient units of the PUK for an RCT. Prior to the first session, patients' electronic files will be screened for inclusion and exclusion criteria and to document medical information, such as current primary diagnoses and current medication. Participants will be randomly assigned to an IRT group or a TAU control group. T0: The first session will consist of informed consent and a first set of self-report questionnaires and interviews, which will assess demographic and personal information, primary psychiatric diagnoses, symptom severity of primary psychiatric diagnoses, psychotherapy motivation and hopefulness, nightmare frequency, nightmare distress, nightmare effects, nightmare content, overall sleep quality, and dream experiences and believes. At the end of the session, both groups will receive a dream diary, which they will fill out for each night for 4 consecutive weeks. The diary will measure nightmare frequency, nightmare distress, nightmare intensity, nightmare content, and if and for how long patients did their imagery exercises.T1: One week later, patients will hand in the completed questionnaires and the IRT group will receive a short IRT intervention. During the IRT session, the therapist will fill out a short questionnaire assessing characteristics of the imagery rescription session. The control group will receive a session in which potential problems with the dream diary will be discussed. Patients in the IRT group will be instructed to use imagery exercises for 10 to 15 minutes a day for the rest of the study period.T2: One week after the IRT or control session, patients will receive self-report questionnaires, which will assess symptom severity of primary psychiatric diagnoses, psychotherapy motivation and hopefulness, nightmare frequency, nightmare distress, nightmare effects, nightmare content, overall sleep quality, and dream experiences and believes. Patients of the IRT group will have the opportunity to ask questions about their treatment. T3: One week later, patients will hand in the completed questionnaires and they will receive the same questionnaires to fill out again. Additionally, patients will receive a questionnaire assessing whether and for how long patients did their imagery exercises during the study period. Patients will also hand in their dream diaries. A week later the questionnaires and dream diaries will be collected. Each patient will receive participant reimbursement of 30 Swiss francs (CHF) for their participation in the study. Furthermore, after data is collected, each patients from the control group will be offered an IRT session.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from the inpatient units at the Psychiatric University Hospital Zurich (PUK) between 18 and 65
* Self-reporting nightmares causing sleep disruption or significant emotional distress
* Currently receiving inpatient care at the PUK
* Fluent in German and able to understand the instructions

Exclusion Criteria:

* No self-reporting nightmares causing sleep disruption or significant emotional distress
* Psychotherapy for nightmare symptoms specifically, currently or in the preceding 12 months
* Not able or willing to engage in imagery exercises
* Patients with a one on one or 15- / 30-minute visual control by the nursing personnel because of risk of suicidal tendencies or the risk of harming others
* Head injury
* Cognitive impairment or other severe symptoms that would interfere with understanding instructions and questionnaires or participation in the study
* Neurological disease
* Shift work
* Trouble speaking and / or understanding the German language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Nightmare frequency (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks
  The Nightmare Frequency Questionnaire and a dream diary will measure the number of nightmares for each night and for each week.
Nightmare distress (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks
  The Nightmare Distress Questionnaire and a dream diary will measure the amount of waking distress associated with nightmares for each night and for each week. Higher Nightmare Distress Questionnaire scores indicate higher nightmare distress (minimum value: 0, maximum value: 52).
Nightmare Intensity (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks
  An adapted version of the Mannheim Dream Questionnaire and a dream diary will measure the intensity of the nightmares of a person (waking up from the nightmare, emotional intensity during the nightmare, how clearly patients remember the nightmare after waking up) for each night and for each week.

SECONDARY OUTCOMES:
Dream experiences and believes (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Mannheim Dream Questionnaire will measure recall of dreams and nightmares, different dream types (nightmares, lucid dreaming), attitude towards dreaming, what dreamers do with their dreams (telling the dream, recording the dream), and effects of dreams on waking life (creative dreams, problem solving dreams, déjà vu experiences based on dreams) for each week.
Overall sleep quality (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Pittsburgh Sleep Quality Index as well as a dream diary will measure the quality of a person's sleep for each night and each week. Higher Pittsburgh Sleep Quality Index scores indicate worse sleep quality (minimum value: 0, maximum value: 21).
Nightmare effects (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Nightmare Effects Survey will measure negative consequences of nightmares on different spheres of life (sleep, work, relationships, daytime energy, school, mood, sex life, diet, mental health, physical health, leisure activities) for each week. Higher Nightmare Effects Survey scores indicate a higher effect of nightmares on daily life (minimum value: 0, maximum value: 44).
Nightmare content (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Mannheim Dream Questionnaire and a dream diary will measure the qualitative content of each nightmare during a subject's participation period.
Severity of depressive symptoms (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Beck Depression Inventory will measure current severity of depressive symptoms (minimum value: 0, maximum value: 63). Higher scores indicate a higher severity.
Severity of anxiety symptoms (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Beck Anxiety Inventory will measure current severity of anxiety symptoms (minimum value: 0, maximum value: 63). Higher scores indicate a higher severity.
Severity of alcohol use (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Alcohol Use Disorders Identification Test will measure current severity of alcohol use (minimum value: 0, maximum value: 40). Higher scores indicate a higher severity.
Severity of drug use (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Drug Use Disorders Identification Test will measure current severity of drug use (minimum value: 0, maximum value: 44). Higher scores indicate a higher severity.
Severity of PTSD symptoms (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The PTSD Checklist for DSM-5 will measure current severity of PTSD symptoms (minimum value: 0, maximum value: 80). Higher scores indicate a higher severity.
Severity of psychotic symptoms (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Community Assessment of Psychic Experiences will measure current severity of psychotic symptoms (frequency and distress score with minimum value: 0, maximum value: 126). Higher scores indicate a higher severity.
Severity of schizophrenia symptoms (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Positive and Negative Syndrom Scale will measure current severity of schizophrenia symptoms (minimum value: 30, maximum value: 210). Higher scores indicate a higher severity.

OTHER OUTCOMES:
Demographic and personal information | Baseline
  A questionnaire will measure demographic and medical background information, such as sex, age, nationality, marital status, residence permit status, children, life situation, highest education, current or last work situation, current social situation, socioeconomic status.
Primary psychiatric diagnosis | Baseline
  The Mini International Neuropsychiatric Interview is a diagnostic interview, which will measure, which psychiatric diagnosis / diagnoses are met according to the International Classification of Diseases (ICD-10) and the Diagnostic and Statistical Manual of Mental Disorders (DSM 4).
Current medication | Baseline, 2 weeks, 3 weeks, 4 weeks
  A medication protocol will document current medication.
Frequency of imagery exercises during the study participation | Baseline, 2 weeks, 3 weeks, 4 weeks
  A questionnaire and a dream diary will ask participants in the IRT group if they did their daily imagery exercises for each day and for the whole study period.
Duration of imagery exercises during the study participation | Baseline, 2 weeks, 3 weeks, 4 weeks
  A questionnaire and a dream diary will ask participants in the IRT group for how long they did their daily imagery exercises for each day and for the whole study period.
Characteristics of the imagery rescription session: Trauma relation of the rescripted nightmare | 1 week after baseline
  A questionnaire, which will be filled out by the therapist during the IRT session, will measure whether the rescripted nightmare is related to a traumatic experience or other aversive life events.
Characteristics of the imagery rescription session: Similarity of the new narrative to the rescripted nightmare | 1 week after baseline
  A questionnaire, which will be filled out by the therapist during the IRT session, will measure how similar the new narrative is to the rescripted nightmare.
Characteristics of the imagery rescription session: Exposure to rescripted nightmare | 1 week after baseline
  A questionnaire, which will be filled out by the therapist during the IRT session, will measure the amount of exposure to the nightmare during the session.
Characteristics of the imagery rescription session: Support by the therapist | 1 week after baseline
  A questionnaire, which will be filled out by the therapist during the IRT session, will measure the amount of support provided by the therapist during the session.
Characteristics of the imagery rescription session: Emotional intensity of the nightmare | 1 week after baseline
  Patients will be asked to rate the emotional intensity of the rescripted nightmare on a scale from 1 to 9.
Characteristics of the imagery rescription session: Emotional intensity of the new narrative | 1 week after baseline
  Patients will be asked to rate the emotional intensity of the rescripted nightmare on a scale from 1 to 9.
Psychotherapy motivation and hopefulness (change from baseline to 1 and 2 weeks after intervention) | Baseline, 2 weeks, 3 weeks, 4 weeks
  The Patient Questionnaire on Therapy Expectation and Evaluation will measure psychotherapy motivation, treatment fit as well as hopefulness of patients regarding their general psychotherapy for each week. Higher scores indicate higher psychotherapy motivation (minimum value: 11, maximum value: 55).

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Psychiatric Association (APA) (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Washington, DC.
- [Background] Eiser AS. Dream disorders and treatment. Curr Treat Options Neurol. 2007 Sep;9(5):317-24. PMID 17716595
- [Background] Ferini-Strambi, L., Fantini, M. L. (2008). Sleep and quality of life in REM sleep parasomnia. In J. C. Verster, S. R. Pandi-Perumal, & D. L. Streiner (Ed.), Sleep and quality of life in clinical medicine (pp. 119-126). New York City: Humana Press.
- [Background] Zadra A, Pilon M, Donderi DC. Variety and intensity of emotions in nightmares and bad dreams. J Nerv Ment Dis. 2006 Apr;194(4):249-54. doi: 10.1097/01.nmd.0000207359.46223.dc. PMID 16614545
- [Background] Levin R, Nielsen TA. Disturbed dreaming, posttraumatic stress disorder, and affect distress: a review and neurocognitive model. Psychol Bull. 2007 May;133(3):482-528. doi: 10.1037/0033-2909.133.3.482. PMID 17469988
- [Background] Sandman N, Valli K, Kronholm E, Revonsuo A, Laatikainen T, Paunio T. Nightmares: risk factors among the Finnish general adult population. Sleep. 2015 Apr 1;38(4):507-14. doi: 10.5665/sleep.4560. PMID 25325474
- [Background] Mume, C. O. (2009). Nightmare in schizophrenic and depressed patients, European Journal of Psychiatry, 23(3), 177-183.
- [Background] Swart ML, van Schagen AM, Lancee J, van den Bout J. Prevalence of nightmare disorder in psychiatric outpatients. Psychother Psychosom. 2013;82(4):267-8. doi: 10.1159/000343590. Epub 2013 Jun 1. No abstract available. PMID 23735876
- [Background] Cernovsky ZZ. MMPI and nightmares in male alcoholics. Percept Mot Skills. 1985 Dec;61(3 Pt 1):841-2. doi: 10.2466/pms.1985.61.3.841. PMID 4088773
- [Background] Cernovsky ZZ. MMPI and nightmare reports in women addicted to alcohol and other drugs. Percept Mot Skills. 1986 Jun;62(3):717-8. doi: 10.2466/pms.1986.62.3.717. PMID 3725511
- [Background] Duke LA, Allen DN, Rozee PD, Bommaritto M. The sensitivity and specificity of flashbacks and nightmares to trauma. J Anxiety Disord. 2008;22(2):319-27. doi: 10.1016/j.janxdis.2007.03.002. Epub 2007 Mar 12. PMID 17434287
- [Background] Krakow B, Schrader R, Tandberg D, Hollifield M, Koss MP, Yau CL, Cheng DT. Nightmare frequency in sexual assault survivors with PTSD. J Anxiety Disord. 2002;16(2):175-90. doi: 10.1016/s0887-6185(02)00093-2. PMID 12194543
- [Background] Reeve S, Sheaves B, Freeman D. Sleep Disorders in Early Psychosis: Incidence, Severity, and Association With Clinical Symptoms. Schizophr Bull. 2019 Mar 7;45(2):287-295. doi: 10.1093/schbul/sby129. PMID 30202909
- [Background] Ellis TE, Rufino KA, Nadorff MR. Treatment of Nightmares in Psychiatric Inpatients With Imagery Rehearsal Therapy: An Open Trial and Case Series. Behav Sleep Med. 2019 Mar-Apr;17(2):112-123. doi: 10.1080/15402002.2017.1299738. Epub 2017 Mar 23. PMID 28332861
- [Background] Nadorff MR, Lambdin KK, Germain A. Pharmacological and non-pharmacological treatments for nightmare disorder. Int Rev Psychiatry. 2014 Apr;26(2):225-36. doi: 10.3109/09540261.2014.888989. PMID 24892897
- [Background] Ohayon MM, Shapiro CM. Sleep disturbances and psychiatric disorders associated with posttraumatic stress disorder in the general population. Compr Psychiatry. 2000 Nov-Dec;41(6):469-78. doi: 10.1053/comp.2000.16568. PMID 11086154
- [Background] Li SX, Zhang B, Li AM, Wing YK. Prevalence and correlates of frequent nightmares: a community-based 2-phase study. Sleep. 2010 Jun;33(6):774-80. doi: 10.1093/sleep/33.6.774. PMID 20550018
- [Background] Nadorff MR, Nadorff DK, Germain A. Nightmares: Under-Reported, Undetected, and Therefore Untreated. J Clin Sleep Med. 2015 Jul 15;11(7):747-50. doi: 10.5664/jcsm.4850. PMID 25845898
- [Background] Kellner R, Neidhardt J, Krakow B, Pathak D. Changes in chronic nightmares after one session of desensitization or rehearsal instructions. Am J Psychiatry. 1992 May;149(5):659-63. doi: 10.1176/ajp.149.5.659. PMID 1349459
- [Background] Aurora RN, Zak RS, Auerbach SH, Casey KR, Chowdhuri S, Karippot A, Maganti RK, Ramar K, Kristo DA, Bista SR, Lamm CI, Morgenthaler TI; Standards of Practice Committee; American Academy of Sleep Medicine. Best practice guide for the treatment of nightmare disorder in adults. J Clin Sleep Med. 2010 Aug 15;6(4):389-401. PMID 20726290
- [Background] Augedal AW, Hansen KS, Kronhaug CR, Harvey AG, Pallesen S. Randomized controlled trials of psychological and pharmacological treatments for nightmares: a meta-analysis. Sleep Med Rev. 2013 Apr;17(2):143-52. doi: 10.1016/j.smrv.2012.06.001. Epub 2012 Oct 6. PMID 23046846
- [Background] Hansen K, Hofling V, Kroner-Borowik T, Stangier U, Steil R. Efficacy of psychological interventions aiming to reduce chronic nightmares: a meta-analysis. Clin Psychol Rev. 2013 Feb;33(1):146-55. doi: 10.1016/j.cpr.2012.10.012. Epub 2012 Nov 7. PMID 23186732
- [Background] Krakow B, Hollifield M, Johnston L, Koss M, Schrader R, Warner TD, Tandberg D, Lauriello J, McBride L, Cutchen L, Cheng D, Emmons S, Germain A, Melendrez D, Sandoval D, Prince H. Imagery rehearsal therapy for chronic nightmares in sexual assault survivors with posttraumatic stress disorder: a randomized controlled trial. JAMA. 2001 Aug 1;286(5):537-45. doi: 10.1001/jama.286.5.537. PMID 11476655
- [Background] Krakow B, Kellner R, Pathak D, Lambert L. Imagery rehearsal treatment for chronic nightmares. Behav Res Ther. 1995 Sep;33(7):837-43. doi: 10.1016/0005-7967(95)00009-m. PMID 7677723
- [Background] Spoormaker VI, Schredl M, van den Bout J. Nightmares: from anxiety symptom to sleep disorder. Sleep Med Rev. 2006 Feb;10(1):19-31. doi: 10.1016/j.smrv.2005.06.001. Epub 2005 Dec 27. PMID 16377217
- [Background] Belicki K. Nightmare frequency versus nightmare distress: relations to psychopathology and cognitive style. J Abnorm Psychol. 1992 Aug;101(3):592-7. doi: 10.1037//0021-843x.101.3.592. PMID 1500619
- [Background] Kales A, Soldatos CR, Caldwell AB, Charney DS, Kales JD, Markel D, Cadieux R. Nightmares: clinical characteristics and personality patterns. Am J Psychiatry. 1980 Oct;137(10):1197-201. doi: 10.1176/ajp.137.10.1197. PMID 7416265
- [Background] Schredl, M. (2003). Continuity between waking and dreaming: A proposal for a mathematical model, Sleep and Hypnosis, 5(1), 26-39.
- [Background] Wood JM, Bootzin RR. The prevalence of nightmares and their independence from anxiety. J Abnorm Psychol. 1990 Feb;99(1):64-8. doi: 10.1037//0021-843x.99.1.64. PMID 2307768
- [Background] Hefez A, Metz L, Lavie P. Long-term effects of extreme situational stress on sleep and dreaming. Am J Psychiatry. 1987 Mar;144(3):344-7. doi: 10.1176/ajp.144.3.344. PMID 3826435
- [Background] Krystal AD, Thakur M, Roth T. Sleep disturbance in psychiatric disorders: effects on function and quality of life in mood disorders, alcoholism, and schizophrenia. Ann Clin Psychiatry. 2008 Jan-Mar;20(1):39-46. doi: 10.1080/10401230701844661. PMID 18297585
- [Background] van Schagen, A., Lancee, J., Spoormaker, V., van den Bout, J. (2016). Long-term treatment effects of Imagery Rehearsal Therapy for nightmares in a population with diverse psychiatric disorders, International Journal of Dream Research, 9, 67-70. doi: 10.11588/ijodr.2016.1.24953.
- [Background] Cukrowicz, K. C., Otamendi, A., Pinto, J. V., Bernert, R. A., Krakow, B., & Joiner, T. E., Jr. (2006). The impact of insomnia and sleep disturbances on depression and suicidality, Dreaming, 16(1), 1-10. doi: 10.1037/1053-0797.16.1.1
- [Background] Sjostrom N, Waern M, Hetta J. Nightmares and sleep disturbances in relation to suicidality in suicide attempters. Sleep. 2007 Jan;30(1):91-5. doi: 10.1093/sleep/30.1.91. PMID 17310869
- [Background] Sjostrom N, Hetta J, Waern M. Persistent nightmares are associated with repeat suicide attempt: a prospective study. Psychiatry Res. 2009 Dec 30;170(2-3):208-11. doi: 10.1016/j.psychres.2008.09.006. Epub 2009 Nov 8. PMID 19900715
- [Background] Tanskanen A, Tuomilehto J, Viinamaki H, Vartiainen E, Lehtonen J, Puska P. Nightmares as predictors of suicide. Sleep. 2001 Nov 1;24(7):844-7. PMID 11683487
- [Background] Germain, A., Krakow, B., Faucher, B., Zadra, A., Nielsen, T., Hollifield, M., Warner, T. D.,& Koss, M. P. (2004). Increased mastery elements associated with imagery rehearsal treatment for nightmares in sexual assault survivors with PTSD, Dreaming, 14(4), 195-206. doi: 10.1037/1053-0797.14.4.195
- [Background] Arntz, A. (2012). Imagery rescripting as a therapeutic technique: Review of clinical trials, basic studies, and research agenda, Journal of Experimental Psychopathology, 3, 189-208. doi: 10.5127/jep.024211
- [Background] Hagenaars MA, Arntz A. Reduced intrusion development after post-trauma imagery rescripting; an experimental study. J Behav Ther Exp Psychiatry. 2012 Jun;43(2):808-14. doi: 10.1016/j.jbtep.2011.09.005. Epub 2011 Sep 21. PMID 22178473
- [Background] Krakow, B. (2004). Imagery Rehearsal Therapy for chronic posttraumatic nightmares: A mind's eye view. In R. I. Rosner, W. J. Lyddon, & A. Freeman (Ed.), Cognitive therapy and dreams (pp. 89-109). New York: Springer Publishing Co.
- [Background] Nappi CM, Drummond SP, Hall JM. Treating nightmares and insomnia in posttraumatic stress disorder: a review of current evidence. Neuropharmacology. 2012 Feb;62(2):576-85. doi: 10.1016/j.neuropharm.2011.02.029. Epub 2011 Mar 17. PMID 21396945
- [Background] Forbes D, Phelps A, McHugh T. Treatment of combat-related nightmares using imagery rehearsal: a pilot study. J Trauma Stress. 2001 Apr;14(2):433-42. doi: 10.1023/A:1011133422340. PMID 11469167
- [Background] Sheaves, B., Onwumere, J., Keen, N., & Kuipers, E. (2015). Treating your worst nightmare: A case-series of Imagery Rehearsal Therapy for nightmares in individuals experiencing psychotic symptoms, The Cognitive Behaviour Therapist, 8(27), 1-17. doi: 10.1017/S1754470X15000665
- [Background] Lu M, Wagner A, Van Male L, Whitehead A, Boehnlein J. Imagery rehearsal therapy for posttraumatic nightmares in U.S. veterans. J Trauma Stress. 2009 Jun;22(3):236-9. doi: 10.1002/jts.20407. PMID 19444882
- [Background] Krakow B, Kellner R, Neidhardt J, Pathak D, Lambert L. Imagery rehearsal treatment of chronic nightmares: with a thirty month follow-up. J Behav Ther Exp Psychiatry. 1993 Dec;24(4):325-30. doi: 10.1016/0005-7916(93)90057-4. PMID 8077451
- [Background] Kunze AE, Arntz A, Morina N, Kindt M, Lancee J. Efficacy of imagery rescripting and imaginal exposure for nightmares: A randomized wait-list controlled trial. Behav Res Ther. 2017 Oct;97:14-25. doi: 10.1016/j.brat.2017.06.005. Epub 2017 Jun 16. PMID 28668770